CLINICAL TRIAL: NCT05579288
Title: Use of Nitrous Oxide for Pain Alleviation in Women Undergoing Osmotic Dilator Insertion for Second Trimester Dilatation and Evacuation
Brief Title: Use of Nitrous Oxide for Pain Alleviation in Women Undergoing Osmotic Dilator Insertion for Dilatation and Evacuation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-22-8935-ST-CTIL
Record Dates: First submitted 2022-09-22; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-04

CONDITIONS: Pain Alleviation; Dilatation and Evacuation; Laminaria Placement; Nitrous Oxide
Keywords: Pain Alleviation; Dilatation and Evacuation; Laminaria Placement; Nitrous Oxide
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Arm (Experimental): Patients will receive inhaled N2O/O2 (70% N2O and 30% O2). A sterile bivalve speculum will be placed. Laminaria will be inserted. Inhaled N2O/O2 will be stopped after speculum removal.
  Interventions: Drug: Nitrous oxide (N2O/O2)
- Control Arm (Placebo Comparator): Patients will receive inhaled O2 (100% O2). A sterile bivalve speculum will be placed. Laminaria will be inserted. Inhaled O2 will be stopped after speculum removal.
  Patients will receive inhaled O2 (100% O2) throughout the procedure until speculum removal.
  Interventions: Drug: Oxygen (O2)

INTERVENTIONS:
Drug: Nitrous oxide (N2O/O2) — Nitrous oxide (N2O/O2) for pain alleviation
  Arms: Study Arm
Drug: Oxygen (O2) — Oxygen (O2) as placebo for control group
  Arms: Control Arm

SUMMARY:
A randomised control study aiming to examine whether inhaled N2O/O2 during cervical preparation for second trimester dilatation and evacuation with osmotic dilators (laminaria) alleviates pain and is superior to placebo.

DETAILED DESCRIPTION:
Introduction:

Women undergoing second trimester abortion often undergo preparation of the cervix prior to the Dilatation and Evacuation (D&E). Women may undergo preparation with osmotic dilators (laminaria) or prostaglandins, both methods are effective and safe for cervical preparation(1). In our institution, the protocol for cervical preparation in the second trimester with osmotic dilator insertion takes place 24 hours before the procedure in the gynecologic emergency room/clinic. Currently, the protocol does not include any method of pain relief during the cervix preparation procedure.

At this time, besides general anesthesia, there are no satisfactory evidence-based methods for pain alleviation for osmotic dilators insertion. For example, a recent randomized controlled trial showed topical application of lidocaine spray to the cervix before insertion did not result in lower reported pain as compared with placebo(2).

Inhaled nitrous oxide administered with oxygen (N2O/O2) is an acceptable, effective and widely used method for pain relief in short painful pediatric ,dental and urologic procedures(3-5), as well as in the labor room and in the emergency room(6, 7). N2O/O2 has analgesic, anxiolytic and amnestic properties. N2O/O2 has rapid onset and reversal with minimal side effects and few contraindications. Side effects of N2O/O2 are relatively minor and include nausea, dizziness, drowsiness, light-headedness, and diaphoresis. Contraindications include congenital heart defects, pulmonary hypertension, megaloblastic anemia and relatively low blood O2 saturation (<95%)(8, 9).

A recent randomized controlled trial showed inhaled N2O/O2 is associated with less pain compared to oral sedation for pain management during in-office hysteroscopic sterilization(9) To the best of our knowledge, there is no literature regarding the efficacy of use of nitrous oxide for pain alleviation in women undergoing osmotic dilator insertion for second trimester Dilatation and Evacuation.

Goal:

To examine whether inhaled N2O/O2 during cervical preparation for second trimester dilatation and evacuation alleviates pain and is superior to placebo.

Methods:

A prospective randomized placebo-controlled trial consisting of two groups:

Inhaled N2O/O2 (group 1) Placebo group (O2 only) (group 2)

Women undergoing dilatation and evacuation in the second trimester and are about to undergo cervical dilatation with osmotic dilators (laminaria) will be invited to participate in a randomized placebo control trial comparing Inhaled N2O/O2 or placebo (O2 only).

The recruitment and trial will take place in the emergency room/clinic where the women come a day before the D&E for cervical preparation. This procedure is routinely performed in a gynecologic chair without any sedation thus assessing pain scores is possible.

Informed consent will be obtained from each participant. Randomization will be performed using a computer randomization generator. After enrollment, patients will be randomized into one of the two study arms. allocation to the two treatment groups will be concealed in sequentially numbered opaque envelopes that will be opened only by the nurse actually administering the gas (either inhaled N2O/O2 or inhaled oxygen). The participant and physician will be completely blinded to the intervention.

Participants will be asked about their most severe pain during menses and asked to rate it from 0 to 10.

The patient will be placed in the lithotomy position.

Group1: Patients will receive inhaled N2O/O2 (70% N2O and 30% O2). A sterile bivalve speculum will be placed. Laminaria will be inserted. Inhaled N2O/O2 will be stopped after speculum removal.

Group2: Patients will receive inhaled O2 (100% O2). A sterile bivalve speculum will be placed. Laminaria will be inserted. Inhaled O2 will be stopped after speculum removal.

Patients will receive inhaled O2 (100% O2) throughout the procedure until speculum removal.

Pain will be assessed at 7-time intervals using a visual analog pain scale 0 (no pain) to 100 (worst possible pain) - 1.Prior to mask application, 2. Before speculum insertion, 3. Immediately after speculum insertion, 4. Immediately after insertion of first laminaria, 5. Immediately after insertion of last laminaria, 6. After speculum removal (including actual VAS and recall of maximal VAS during the procedure), 7. Before the D&E the next day.

Satisfaction with the procedure will be collected as well- overall satisfaction (0-100) and satisfaction with pain control (0-100).

Data regarding adverse events will be collected as well.

Primary outcome:

Self-report of pain score immediately following speculum removal.

Secondary outcome:

Self-report of maximal pain during the procedure.

The protocol will not be repeated if a participant is to return for further laminaria insertion.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent

Exclusion Criteria:

* D&E due to PPROM or infection.
* Known N2O allergy.
* Contraindication to N2O use - Congenital heart defects, pulmonary hypertension, megaloblastic anemia, O2 blood saturation <95%

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Self-report of change in pain score immediately following speculum removal | 2 days
  Pain will be assessed at 7-time intervals using a visual analog pain scale 0 (no pain) to 100 (worst possible pain) - 1.Prior to mask application, 2. Before speculum insertion, 3. Immediately after speculum insertion, 4. Immediately after insertion of first laminaria, 5. Immediately after insertion of last laminaria, 6. After speculum removal (including actual VAS and recall of maximal VAS during the procedure), 7. Before the D&E the next day.

SECONDARY OUTCOMES:
Self-report of change in maximal pain during the procedure | 2 days
  Pain will be assessed at 7-time intervals using a visual analog pain scale 0 (no pain) to 100 (worst possible pain) - 1.Prior to mask application, 2. Before speculum insertion, 3. Immediately after speculum insertion, 4. Immediately after insertion of first laminaria, 5. Immediately after insertion of last laminaria, 6. After speculum removal (including actual VAS and recall of maximal VAS during the procedure), 7. Before the D&E the next day.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newmann SJ, Dalve-Endres A, Diedrich JT, Steinauer JE, Meckstroth K, Drey EA. Cervical preparation for second trimester dilation and evacuation. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007310. doi: 10.1002/14651858.CD007310.pub2. PMID 20687085
- [Background] Meyer R, Cahan T, Yagel I, Afek A, Derazne E, Bar-Shavit Y, Yuval Y, Admon D, Shina A. A double-blind randomized trial comparing lidocaine spray and placebo spray anesthesia prior to cervical laminaria insertion. Contraception. 2020 Nov;102(5):332-338. doi: 10.1016/j.contraception.2020.07.002. Epub 2020 Jul 8. PMID 32652092
- [Background] Wood M. The safety and efficacy of intranasal midazolam sedation combined with inhalation sedation with nitrous oxide and oxygen in paediatric dental patients as an alternative to general anaesthesia. SAAD Dig. 2010 Jan;26:12-22. PMID 20151606
- [Background] Burnweit C, Diana-Zerpa JA, Nahmad MH, Lankau CA, Weinberger M, Malvezzi L, Smith L, Shapiro T, Thayer K. Nitrous oxide analgesia for minor pediatric surgical procedures: an effective alternative to conscious sedation? J Pediatr Surg. 2004 Mar;39(3):495-9; discussion 495-9. doi: 10.1016/j.jpedsurg.2003.11.037. PMID 15017577
- [Background] Young A, Ismail M, Papatsoris AG, Barua JM, Calleary JG, Masood J. Entonox(R) inhalation to reduce pain in common diagnostic and therapeutic outpatient urological procedures: a review of the evidence. Ann R Coll Surg Engl. 2012 Jan;94(1):8-11. doi: 10.1308/003588412X13171221499702. PMID 22524905
- [Background] Broughton K, Clark AG, Ray AP. Nitrous Oxide for Labor Analgesia: What We Know to Date. Ochsner J. 2020 Winter;20(4):419-421. doi: 10.31486/toj.19.0102. PMID 33408580
- [Background] Descamps MJ, Gwilym S, Weldon D, Holloway V. Prospective audit of emergency department transit times associated with entonox analgesia for reduction of the acute, traumatic dislocated shoulder. Accid Emerg Nurs. 2007 Oct;15(4):223-7. doi: 10.1016/j.aaen.2007.07.008. Epub 2007 Oct 29. PMID 17911025
- [Background] O'Sullivan I, Benger J. Nitrous oxide in emergency medicine. Emerg Med J. 2003 May;20(3):214-7. doi: 10.1136/emj.20.3.214. PMID 12748131
- [Background] Schneider EN, Riley R, Espey E, Mishra SI, Singh RH. Nitrous oxide for pain management during in-office hysteroscopic sterilization: a randomized controlled trial. Contraception. 2017 Mar;95(3):239-244. doi: 10.1016/j.contraception.2016.09.006. Epub 2016 Sep 9. PMID 27621048
- [Background] Mercier RJ, Liberty A. Intrauterine lidocaine for pain control during laminaria insertion: a randomized controlled trial. Contraception. 2014 Dec;90(6):594-600. doi: 10.1016/j.contraception.2014.07.008. Epub 2014 Jul 23. PMID 25139724